CLINICAL TRIAL: NCT07269093
Title: Efficacy in Preventing Hypertrophic Scars: A Randomised Controlled Trial Comparing Chitosan Cream, Silicone Gel & Olive Oil
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Esther Tan Hui Min, Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: USM/JEPeM/KK/25060539
Record Dates: First submitted 2025-11-21; First posted 2025-12-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hypertrophic Scars
Keywords: Chitosan; silicone gel; olive oil; hypertrophic scars; prevention
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silicone gel (Active Comparator): Silicone gel application twice a day for 8 weeks
  Interventions: Device: Silicone Gel
- Chitosan cream (Experimental): Chitosan cream application twice a day for 8 weeks
  Interventions: Device: Chitosan cream
- Olive oil (Placebo Comparator): Olive oil application twice a day for 8 weeks
  Interventions: Device: Olive Oil Topical Oil

INTERVENTIONS:
Device: Chitosan cream — Application of Chitosan cream twice daily for 8 weeks
  Arms: Chitosan cream
Device: Silicone Gel — Application of silicone gel twice a day for 8 weeks
  Arms: Silicone gel
Device: Olive Oil Topical Oil — Application of olive oil twice daily for 8 weeks
  Arms: Olive oil

SUMMARY:
The goal of this clinical trial is to compare the efficacy of three different topical applications in preventing hypertrophic scars in adults with scars healed after suturing. The main question it aims to answer is: Is Chitosan cream effective in preventing hypertrophic scars?

Researchers will compare Chitosan cream with silicone gel and olive oil to see if there is any difference in their efficacies.

Participants will be randomly assigned to three groups, with each group using a different topical application. They will be instructed to:

* apply the topical application on their scar twice a day for 8 weeks
* attend follow-up visits at 4, 12 and 24 weeks for a doctor to assess their scar and take clinical photographs
* immediately inform the researcher if they experience any side effects

DETAILED DESCRIPTION:
This is a 3-arm single-blinded randomised controlled trial to study the efficacy of three topical applications in preventing hypertrophic scars. The general objective is to investigate the efficacy of Chitosan cream in preventing hypertrophic scars compared to other topical applications commonly used; silicone gel and olive oil. The hypothesis is that Chitosan cream shows comparable efficacy in preventing hypertrophic scars compared to silicone gel and olive oil.

The study population consists of patients who had traumatic or surgical scars that have healed by primary intention in the Unit of Reconstructive Sciences, Hospital Pakar USM, Plastic & Reconstructive Surgery Unit of Hospital Raja Perempuan Zainab II and the Plastic & Reconstructive Surgery Department of Hospital Kuala Lumpur and have met the study inclusion criteria.

Patients who meet the inclusion criteria will be given a topical application (Chitosan cream / silicone gel / olive oil) which is assigned randomly by computer software (SPSS version 29). The topical applications is to be applied twice daily from the 14th day since wounding. The investigator will be blinded to the topical application given to the patient. Both patient and investigator will assess the scar using Patient & Observer Scar Assessment Scale (POSAS) version 3.0 and scars will be photographed under fixed camera settings & lighting conditions. Patients will come for follow-up on weeks 4, 12 & 24 and the scar assessment will be repeated by both patient & the same observer. Serial photographs will also be taken each visit. At the end of the 24 weeks, photographs of the scars will be reviewed by three independent plastic surgeons and scored using the Scar Cosmesis & Assessment Rating (SCAR) Scale. Both the scores from the clinical & photographic scar assessments will be evaluated to compare the efficacy of each topical application. The duration of the study is from Nov 2025-Nov 2026.

ELIGIBILITY:
Inclusion Criteria:

* Patients with traumatic or surgical wounds which have healed by primary intention within 14 days
* Length of scar at least 3cm

Exclusion Criteria:

* Patients with seafood allergy
* Patients with scar from wounds that were complicated by infection or wound breakdown
* Patients who have undergone scar treatment by other modalities
* Patients with history of keloids / hypertrophic scars
* Pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) scores | Enrolment to 24 weeks
  Each item is rated on a 5-point score. The lowest score is '1' which corresponds to the situation of normal skin. Score '5' being the largest difference from normal skin.
Scar Assessment and Rating (SCAR) Scale scores | Enrolment to 24 weeks
  Scores of clinical photographs of each scar by 3 plastic surgeons. Score '0' indicates conditions closest to normal skin. Maximum scores for each item range from 1 to 4, where higher scores indicate larger differences from normal skin.

SECONDARY OUTCOMES:
Side effects | Enrolment to 24 weeks
  Patients are to report any side effects that they experience with use of any topical application. Side effects encountered are recorded.

CONTACTS AND LOCATIONS:
Locations (3):
- Malaysia (3):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Pakar Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No
Patient privacy protection

REFERENCES:
- [Background] Kantor J. Reliability and Photographic Equivalency of the Scar Cosmesis Assessment and Rating (SCAR) Scale, an Outcome Measure for Postoperative Scars. JAMA Dermatol. 2017 Jan 1;153(1):55-60. doi: 10.1001/jamadermatol.2016.3757. PMID 27806156
- [Background] Carriere ME, Mokkink LB, Tyack Z, Westerman MJ, Pijpe A, Pleat J, van de Kar AL, Brown J, de Vet HCW, van Zuijlen PPM. Development of the Patient Scale of the Patient and Observer Scar Assessment Scale (POSAS) 3.0: a qualitative study. Qual Life Res. 2023 Feb;32(2):583-592. doi: 10.1007/s11136-022-03244-6. Epub 2022 Nov 10. PMID 36355319